CLINICAL TRIAL: NCT05989048
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Zavegepant Intranasal (IN) for the Acute Treatment of Migraine in Asian Adults
Brief Title: A Study to Learn About Zavegepant as the Acute Treatment of Migraine in Asian Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C5301008; NCT05989048 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zavegepant (Experimental): Zavegepant intranasal 10 mg
  Interventions: Drug: Zavegepant
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zavegepant — The participants will receive single active dose sufficient to treat 1 migraine headache of moderate or severe intensity within Treatment Phase.
  Arms: Zavegepant
Drug: Placebo — Single dose of matching placebo taken within Treatment Phase.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn how safe and effective zavegepant is compared to placebo in the acute treatment of migraine in Asian adults. Migraine is a very painful headache with other associated symptoms such as nausea, photophobia and phonophobia. A placebo is a harmless treatment that has no medical effect.

This study is seeking for participants who:

* have at least 1 year of migraine history before entering the study.
* have 2 to 8 migraine headache attacks of moderate or severe intensity in each of the 3 months before entering the study.
* have less than 15 days with headaches in each of the 3 months before entering the study. The headaches could be either due to migraine or not.

The participants in this study will receive zavegepant or placebo through intranasal route. Intranasal means medicine which is given through nose. Zavegepant or placebo will be taken if the participants have a migraine headache of moderate or severe intensity.

The study will compare the experiences of people receiving zavegepant to those of the people receiving placebo. This will help see if zavegepant is safe and effective in Asian adults.

Participants will be in this study for up to about 16 weeks. Participants will have 3 study visits at the study clinic and 1 through telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Asian participants aged 18 years or older at screening.
* Participants with minimum 1 year history of migraine (with or without aura) prior to the Screening Visit, consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, including the following:

  1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age.
  2. Migraine attacks, on average, lasting about 4-72 hours if untreated.
  3. Not more than 8 attacks of moderate or severe pain intensity per month within last 3 months.
  4. Participants must be able to distinguish migraine attacks from tension/cluster headaches.
  5. At least 2 consistent migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and throughout the Screening Phase (participant self-report).
  6. Less than 15 days with headaches (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and throughout the Screening Phase (participant self-report).
  7. Participants on prophylactic migraine medication are permitted to remain on therapy if they have been on a stable dose for at least 3 months prior to Screening Visit, and if the dose is not expected to change through the End of Treatment Visit.
  8. Participants with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Exclusion Criteria:

* History of retinal migraine, basilar migraine or hemiplegic migraine.
* History or current evidence of uncontrolled, unstable or recently diagnosed cardiovascular or cardiometabolic disease.
* Major depressive disorder, anxiety disorder, or other significant psychiatric disorder.
* Acute or chronic pain syndromes, psychiatric conditions, dementia, or significant neurological disorders (other than migraine) that interfere with study assessments.
* Conditions that may affect the administration or absorption of the nasal product.
* Medication overuse headaches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1414 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with pain freedom at 2 hours post dose. | 2 hours post dose
  To compare the efficacy of zavegepant with placebo in the acute treatment of migraine by measuring freedom from pain.
Percentage of participants with an MBS (most bothersome symptom) reported before dosing that is absent at 2 hours post dose. | 2 hours post dose
  To compare the efficacy of zavegepant with placebo in the acute treatment of migraine by measuring freedom from MBS.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- China (45):
  - The Second People's hospital of Hefei, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Hainan General Hospital, Haikou, Hainan
  - Renmin Hospital Of Wuhan University, Wuhan, Hebei
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Wuhan Third Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - General Hospital of Ningxia Medical Hospital, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People' Hospital, Xi'an, Shaanxi
  - Xian Gaoxin Hospital, Xi'an, Shaanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng people's Hospital, Liaocheng, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - People's Hospital of Rizhao, Rizhao, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ruian People's Hospital, Rui’an, Zhejiang
  - The First Affiliated Hosptial of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Chongqing University Three Gorges Hospital, Chongqing
  - The fourth people's hospital of chongqing, Chongqing
  - Shanghai East Hospital, Shanghai
  - Tianjin Union Medical Center, Tianjin
- South Korea (12):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inje University - Ilsan Paik Hospital, Goyang-si, Kyǒnggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si, Kyǒnggi-do
  - Dong-A University Hospital, Busan, Pusan-kwangyǒkshi
  - Nowon Eulji Medical Center, Eulji University, Seoul, Seoul-teukbyeolsi [seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Seoul Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kangbuk Samsung Hospital, Seoul
- Taiwan (3):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5301008